CLINICAL TRIAL: NCT01755975
Title: A Phase Ib/IIa Study of Romidepsin in Combination With Lenalidomide in Adults With Relapsed or Refractory Lymphomas and Myeloma
Brief Title: Romidepsin in Combination With Lenalidomide in Adults With Relapsed or Refractory Lymphomas and Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: St. Francis Hospital & Medical Center, Hartford CT (Other); Weill Medical College of Cornell University (Other); University of Nebraska (Other); Celgene Corporation (Industry); Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-170
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; Non-Hodgkin's Lymphoma
Keywords: LENALIDOMIDE (CC-5013); Romidepsin (Istodax); 12-170
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — romidepsin; Lenalidomide

ARMS (1):
- Romidepsin and Lenalidomide (Experimental): This will be a multicentered, open label, phase Ib/IIa trial of romidepsin and lenalidomide in patients with relapsed or refractory lymphomas or multiple myeloma. Lenalidomide will be provided in accordance with the Celgene Corporation's Revlimid REMS® program. Per standard Revlimid REMS® program requirements, all physicians who prescribe lenalidomide for research subjects enrolled into this trial, and all research subjects enrolled into this trial, must be registered in, and must comply with, all requirements of the Revlimid REMS® program. Only enough lenalidomide for one cycle of therapy will be supplied to the patient each cycle.
  Interventions: Drug: Romidepsin; Drug: Lenalidomide

INTERVENTIONS:
Drug: Romidepsin — Romidepsin will be administered intravenously on days 1, 8, and 15 of a 28-day cycle.
Drug: Lenalidomide — Lenalidomide will be taken orally daily for 21 days of a 28-day cycle.

SUMMARY:
The treatments used to treat lymphoma and multiple myeloma sometimes do not always work well or they may only work for a short period of time. This is why new treatments are being tested.

This study will test a new combination of two drugs that are already approved by the Food and Drug Administration for treatment of certain kinds of blood cancers. These drugs are romidepsin and lenalidomide. Both these drugs by themselves have been used to treat lymphoma or multiple myeloma. However, while these drugs are routinely used alone, this is the first time they will be tested together. The mechanism of action of both drugs is not well understood but both have been shown to to be effective by themselves in lymphoma and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed lymphoma or multiple myeloma
* Hodgkin lymphoma is eligible for either phase and will be considered a B-cell lymphoma in the phase IIa study.
* Phase IIa portion, subjects must have B-cell lymphoma, T-cell lymphoma, or multiple myeloma.
* Relapse or progression after at least 1 systemic therapy.
* Measurable disease for phase IIa portion only.
* Lymphoma (includes CTCL patients who are NED in skin): CT or PET/CT by modified Cheson criteria with incorporation of PET.
* Multiple myeloma:.Patient must have measurable disease and therefore must have at least one of the following:

  i. Serum M-protein ≥0.5gm/dL (≥5gm/L) ii. Urine M-protein ≥200mg/24hr iii. Serum FLC assay: involved FLC ≥10mg/dL (≥100mg/L) provided serum FLC ratio is abnormal.
* CTCL: mSWAT >0, or absolute Sezary count ≥ 1000 cells/μL.
* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Previous systemic anti-cancer therapy must have been discontinued at least 3 weeks prior to treatment in this study. If there is progression of disease on that therapy and all adverse effects have resolved to Grade 1 or baseline, in which case 2 weeks is acceptable.
* Previous radiation, hormonal therapy, and surgery must have been discontinued or completed at least 2 weeks prior to treatment in this study and adverse effects must have resolved. Lymph node or other diagnostic biopsy within 2 weeks is not considered exclusionary.
* Short course systemic corticosteroids for disease control, improvement of performance status or non-cancer indication (< 7 days) must have been discontinued at least 7 days prior to study treatment. Stable ongoing corticosteroid use (≥ 30 days) up to an equivalent dose of 15 mg of prednisone is permissible.
* ECOG performance status of ≤ 2 at study entry
* Laboratory test results within these ranges:
* Absolute neutrophil count ≥ 1.0/mm³.
* Platelet count ≥ 70 K/μL, if thrombocytopenia is due to bone marrow involvement platelet count must be ≥ 50 K/μL.
* Renal function assessed by calculated creatinine clearance as follows
* Phase Ib subjects must have calculated creatinine clearance ≥ 50ml/min by Cockcroft-Gault formula.
* Phase IIa subjects must have calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance < 60ml/min and ≥ 30ml/min.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN); 3 x ULN if due to hepatic involvement.
* AST (SGOT) and ALT (SGPT) ≤ 3 x ULN; 5 x ULN if due to hepatic involvement.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix C: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods. † A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Patients who have a standard curative option for their lymphoid malignancy at current state of disease are excluded. For eligibility on this trial, allogeneic stem cell transplantation is not to be considered a standard curative option.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.

Pregnant females. (Lactating females must agree not to breast feed while taking lenalidomide or romidepsin).

* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Prior use of lenalidomide if discontinued due to toxicity.
* Prior therapy with romidepsin if discontinued due to toxicity.
* Concurrent use of other anti-cancer agents or treatments.
* Known seropositive and requiring anti-viral therapy for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Active concurrent malignancy requiring active therapy.
* Known central nervous system or meningeal involvement (in the absence of symptoms investigation into central nervous system involvement is not required). Patients with HTLV1 ATLL and controlled CNS or meningeal involvement may be enrolled after discussion with the MSK principal investigator.
* The following known cardiac abnormalities:
* Congenital long QT syndrome.
* QTc interval ≥ 480 milliseconds
* A QTc interval between 480-499 msec in the presence of a bundle branch block (BBB) or pacemaker is are eligible in phase IIa after discussion with the MSK principal investigator
* Myocardial infarction within 6 months of cycle one, day one (C1D1). Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate.
* Other significant ECG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block. Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Appendix D). In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix E) and/or ejection fraction <45% by MUGA, echocardiogram, or cardiac MRI.
* A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD). Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes.
* Uncontrolled hypertension, i.e., blood pressure (BP) of ≥170/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
* Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* Patients taking drugs leading to significant QTc prolongation unless able to be switched to non-QTc prolonging medication without risk of worsening underlying condition and meet all other inclusion criteria: Medications That May Cause QTc Prolongation).
* Concomitant use of significant CYP3A4 inhibitors unless able to be switched to a non-CYP3A4 inhibiting medication without risk of worsening underlying condition and able to meet all other inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-12; Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Saint Francis/Mount Sinai Regional Cancer Center, Hartford, Connecticut
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level -1: Romidepsin 8 mg/m^2/Lenalidomide 10 mg
- Dose Level 1: Romidepsin 8 mg/m^2/Lenalidomide 15 mg
- Dose Level 2: Romidepsin 8 mg/m^2/Lenalidomide 25 mg
- Dose Level 3: Romidepsin 10 mg/m^2/Lenalidomide 25 mg
- Dose Level 4: Romidepsin 14 mg/m^2/Lenalidomide 25 mg
Period: Overall Study
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 0 | 3 | 7 | 3 | 36
Completed | 0 | 3 | 6 | 3 | 34
Not Completed | 0 | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: No participants accrued to Dose Level -1
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36 | 49
Age, Continuous [Median (Full Range); unit: years] |  | 69 [67 to 72] | 53 [25 to 65] | 53 [38 to 76] | 63 [33 to 84] | 65 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 6 | 2 | 14 | 23
  Male |  | 2 | 1 | 1 | 22 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino |  | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 3 | 7 | 3 | 36 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 2 | 0 | 8 | 10
  Asian |  | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 1 | 1
  Black or African American |  | 0 | 0 | 0 | 0 | 0
  White |  | 3 | 4 | 2 | 23 | 32
  More than one race |  | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 1 | 1 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 3 | 7 | 3 | 36 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities/DLTs
Description: The phase Ib portion of the study is designed to determine the MTD of romidepsin and lenalidomide.
Time Frame: 1 year
Population: No participants treated on Dose Level -1
Measure: Number; unit: DLT's
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36
DLT's |  | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants Evaluable for AEs
Description: Subjects will be evaluated for AEs at each visit with the NCI CTCAE v4.0 used as a guide for the grading of severity.
Time Frame: 1 year
Population: No participants treated on Dose Level -1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36
Participants
  Evaluable for AEs | 0 | 3 | 6 | 3 | 36
  Not Evaluable for AEs | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Assess the Overall Response Rate (ORR)
Description: Overall response rate (ORR), complete response rate, very good partial response/partial response rate will be summarized using proportions and confidence intervals will be provided. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: No participants treated on Dose Level -1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36
Participants
  complete response rate, very good partial response/partial response rate |  | 2 | 3 | 0 | 17
  Stable response or progression of disease |  | 1 | 4 | 3 | 19

4. Secondary Outcome: Complete Response Rate/CRR
Description: CRR is defined as Complete Response Rate. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: No participants treated on Dose Level -1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36
Participants
  Complete Response |  | 1 | 1 | 0 | 6
  No Complete Response |  | 2 | 6 | 3 | 30

5. Secondary Outcome: Assess the Time to Best Response (TTBR)
Description: Duration of response (DOR), and event free survival (EFS). Time to response,duration of response and event free survival will be analyzed by routine survival analysis tools such as Kaplan-Meier estimation or competing risks method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 50 months
Population: No participants treated on Dose Level -1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 3 | 7 | 3 | 36
months
  Progression Free Survival/PFS |  | 5.7 [3.7 to 16.7] | 5.7 [3.7 to 16.7] | 5.7 [3.7 to 16.7] | 5.7 [3.7 to 16.7]
  Overall Survival/OS |  | 24.0 [10.0 to 48.8] | 24.0 [10.0 to 48.8] | 24.0 [10.0 to 48.8] | 24.0 [10.0 to 48.8]
  Duration of Response/DOR |  | 15.7 [4.1 to 26.2] | 15.7 [4.1 to 26.2] | 15.7 [4.1 to 26.2] | 15.7 [4.1 to 26.2]
  Time To Best Response/TTBR |  | 3.7 [1.9 to 9.0] | 3.7 [1.9 to 9.0] | 3.7 [1.9 to 9.0] | 3.7 [1.9 to 9.0]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 5 years, Adverse Events monitored/assessed up to 1 year
Description: No participants treated on Dose Level -1
Groups:
- Dose Level 2: Romidepsin 8 mg/m^2/Lenalidomide 25
Arm/Group | Dose Level -1 | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/3 | 6/7 | 1/3 | 21/36
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 7/7 | 1/3 | 36/36
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 7/7 | 3/3 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level -1 (N=0) | Dose Level 1 (N=3) | Dose Level 2 (N=7) | Dose Level 3 (N=3) | Dose Level 4 (N=36)
Abdominal distension (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | NA | 0 | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | NA | 0 | 2 | 0 | 4
Ankle fracture (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | NA | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | NA | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | NA | 0 | 2 | 0 | 0
Confusion (Psychiatric disorders) | NA | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | 3
Diarrhea (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 1 | 0 | 4
Edema limbs (General disorders) | NA | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
Fatigue (General disorders) | NA | 0 | 2 | 0 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 | 1 | 0 | 2
Fever (General disorders) | NA | 0 | 3 | 0 | 4
Gastrointestinal disorders - Gastroenteritis (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 7
Hypotension (Vascular disorders) | NA | 0 | 0 | 0 | 1
INR increased (Investigations) | NA | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | NA | 1 | 0 | 0 | 3
Mucosal infection (Infections and infestations) | NA | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | NA | 0 | 1 | 0 | 4
Pericardial effusion (Cardiac disorders) | NA | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | NA | 0 | 1 | 0 | 5
Pleural infection (Infections and infestations) | NA | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | NA | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 2
Rhinitis infective (Infections and infestations) | NA | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | NA | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | NA | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | NA | 0 | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | NA | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | NA | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level -1 (N=0) | Dose Level 1 (N=3) | Dose Level 2 (N=7) | Dose Level 3 (N=3) | Dose Level 4 (N=36)
Abdominal pain (Gastrointestinal disorders) | NA | 1 | 1 | 1 | 10
Acute kidney injury (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | NA | 0 | 3 | 0 | 2
Alkaline phosphatase increased (Investigations) | NA | 0 | 1 | 1 | 8
Allergic reaction (Immune system disorders) | NA | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | NA | 1 | 1 | 1 | 5
Anemia (Blood and lymphatic system disorders) | NA | 0 | 7 | 3 | 36
Ankle fracture (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | NA | 1 | 3 | 0 | 28
Anxiety (Psychiatric disorders) | NA | 0 | 0 | 0 | 2
Appendicitis (Infections and infestations) | NA | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | NA | 0 | 1 | 0 | 7
Atrial fibrillation (Cardiac disorders) | NA | 0 | 0 | 0 | 1
Autoimmune disorder (Immune system disorders) | NA | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 3
Bladder infection (Infections and infestations) | NA | 0 | 0 | 0 | 2
Bloating (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | NA | 0 | 7 | 0 | 3
Blurred vision (Eye disorders) | NA | 1 | 0 | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | NA | 0 | 0 | 0 | 2
Chest pain - cardiac (Cardiac disorders) | NA | 0 | 0 | 1 | 0
Chills (General disorders) | NA | 0 | 0 | 0 | 2
Cognitive disturbance (Nervous system disorders) | NA | 0 | 0 | 0 | 2
Concentration impairment (Nervous system disorders) | NA | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | NA | 0 | 3 | 2 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 3 | 1 | 1 | 15
Creatinine increased (Investigations) | NA | 0 | 1 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | NA | 1 | 1 | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | NA | 3 | 4 | 0 | 33
Dizziness (Nervous system disorders) | NA | 0 | 0 | 1 | 11
Dry eye (Eye disorders) | NA | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | NA | 0 | 0 | 1 | 2
Dry skin (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 6
Dysesthesia (Nervous system disorders) | NA | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | NA | 2 | 3 | 3 | 36
Dyspepsia (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 2 | 0 | 16
Edema (General disorders) | NA | 0 | 0 | 0 | 1
Edema face (General disorders) | NA | 0 | 0 | 0 | 1
Edema limbs (General disorders) | NA | 1 | 0 | 0 | 10
Ejection fraction decreased (Investigations) | NA | 0 | 0 | 0 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | NA | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 4
Excess Salivation (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | NA | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | NA | 0 | 0 | 0 | 1
Fatigue (General disorders) | NA | 3 | 1 | 3 | 36
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 | 1 | 0 | 2
Fever (General disorders) | NA | 1 | 7 | 0 | 11
Flatulence (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | NA | 0 | 0 | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Genital edema (Reproductive system and breast disorders) | NA | 0 | 0 | 0 | 2
Glaucoma (Eye disorders) | NA | 0 | 0 | 1 | 0
Gum infection (Infections and infestations) | NA | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | NA | 0 | 1 | 2 | 5
Hearing impaired (Ear and labyrinth disorders) | NA | 0 | 0 | 1 | 1
Hematuria (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 12
Hyperglycemia (Metabolism and nutrition disorders) | NA | 0 | 7 | 0 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 7
Hypermagnesemia (Metabolism and nutrition disorders) | NA | 3 | 7 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | NA | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | NA | 0 | 0 | 1 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 1 | 9
Hypocalcemia (Metabolism and nutrition disorders) | NA | 0 | 4 | 0 | 25
Hypoglycemia (Metabolism and nutrition disorders) | NA | 0 | 7 | 0 | 10
Hypoglycemia (Metabolism and nutrition disorders) | NA | 0 | 2 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | NA | 1 | 5 | 0 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | NA | 0 | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | NA | 0 | 0 | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | NA | 0 | 7 | 0 | 36
Hypothyroidism (Endocrine disorders) | NA | 0 | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | NA | 0 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | NA | 0 | 0 | 2 | 0
Injection site reaction (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
INR increased (Investigations) | NA | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | NA | 2 | 0 | 0 | 4
Leg Cramps (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | NA | 0 | 0 | 0 | 1
Lipase increased (Investigations) | NA | 0 | 2 | 0 | 0
Lung infection (Infections and infestations) | NA | 1 | 2 | 0 | 2
Lymph gland infection (Infections and infestations) | NA | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | NA | 3 | 7 | 3 | 36
Malaise (General disorders) | NA | 0 | 0 | 0 | 3
Middle ear inflammation (Ear and labyrinth disorders) | NA | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 3 | 1 | 0 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 1 | 1 | 7
Nausea (Gastrointestinal disorders) | NA | 2 | 2 | 1 | 36
Neck pain (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 3
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | NA | 3 | 7 | 3 | 36
Night Sweats (Skin and subcutaneous tissue disorders) | NA | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | NA | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | NA | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | NA | 1 | 0 | 1 | 0
Pain (General disorders) | NA | 0 | 0 | 0 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Pain-Shoulder (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | NA | 0 | 0 | 0 | 3
Paresthesia (Nervous system disorders) | NA | 0 | 0 | 0 | 3
Pericardial effusion (Cardiac disorders) | NA | 0 | 0 | 0 | 1
Periorbital edema (Eye disorders) | NA | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | NA | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | NA | 2 | 0 | 0 | 14
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | NA | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | NA | 3 | 7 | 3 | 36
Presyncope (Nervous system disorders) | NA | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | NA | 2 | 0 | 1 | 14
QTc Prolongation (Investigations) | NA | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 11
Rectal pain (Gastrointestinal disorders) | NA | 0 | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | NA | 0 | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | NA | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | NA | 0 | 0 | 0 | 1
Serum amylase increased (Investigations) | NA | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | NA | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | NA | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | NA | 0 | 0 | 0 | 2
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | NA | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | NA | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | NA | 1 | 0 | 1 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | NA | 0 | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | 1 | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | NA | 0 | 1 | 0 | 2
Thromboembolic event (Vascular disorders) | NA | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | NA | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | NA | 2 | 0 | 0 | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | NA | 0 | 1 | 0 | 1
Urinary frequency (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | NA | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | NA | 0 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | NA | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | NA | 3 | 2 | 0 | 18
Watering eyes (Eye disorders) | NA | 1 | 0 | 0 | 3
Weight gain (Investigations) | NA | 0 | 0 | 0 | 2
Weight loss (Investigations) | NA | 3 | 3 | 0 | 13
Wheezing (Respiratory, thoracic and mediastinal disorders) | NA | 2 | 0 | 0 | 1
White blood cell decreased (Investigations) | NA | 1 | 7 | 2 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT01755975/Prot_SAP_000.pdf